CLINICAL TRIAL: NCT00301626
Title: ROSCAP: Reduction of Smoking in Cardiac Patients Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health (NIH) (NIH)
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DA13333-02
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2005-04

CONDITIONS: Nicotine Dependence; Tobacco Dependence; Cardiac Disease
Keywords: tobacco; nicotine; smoking reduction
MeSH Terms: conditions — Tobacco Use Disorder; Heart Diseases; Smoking Reduction

INTERVENTIONS:
Behavioral: smoking reduction intervention (including NRT)

SUMMARY:
Background. The ROSCAP Study was a randomized controlled trial in heart disease patients to test the effect of a smoking reduction intervention on cigarettes per day (cpd) and biochemical and clinical indicators of tobacco exposure. .

ELIGIBILITY:
Inclusion Criteria:

* smoked at least 15 cigarettes per day and had one of 11 cardiovascular disorders: history of myocardial infarction, coronary artery bypass surgery, angioplasty, stent placement, thrombolytic therapy, angina, arrhythmia, a history of cardiac arrest, greater than 50% coronary artery stenosis by angiography, ischemia on exercise tolerance testing or congestive heart failure, required to confirm that they were unwilling or uninterested in setting a stop smoking date in the next 30 days.

Exclusion Criteria:

* 1) unstable angina within the past 2 weeks, 2) unstable psychiatric or substance use disorders or 3) contraindications to nicotine replacement therapy (including pregnancy or intention to become pregnant)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2000-10; Study Completion 2005-01

PRIMARY OUTCOMES:
Smoking reduction

SECONDARY OUTCOMES:
Smoking cessation, biomarker measures

CONTACTS AND LOCATIONS:
Overall Officials: Anne Joseph, MD, MPH, Principal Investigator — Minneapolis VAMC & University of Minnesota
Locations (1):
- Minneapolis VAMC (111-0), Minneapolis, Minnesota, United States